CLINICAL TRIAL: NCT04311918
Title: The Effect of Fluids Flushed in Pediatric Cardiac Catheterization Procedures on Lung Ultrasound Score: A Prospective Observational Study
Brief Title: The Effect of Fluids Flushed in Pediatric Cardiac Catheterization Procedures on Lung Ultrasound Score
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Madkour, Associate professor, Cairo University
Other Study IDs: MD-20-2020
Record Dates: First submitted 2020-03-11; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Congenital Heart Disease
Keywords: congenital - cardiac catheterization
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Therapeutic catheterizations substituted many traditional surgical procedures with the advance of transcatheter techniques.

Pediatric patients are more liable to fluid overload due to their smaller weights compared to adults and the risk increases in pediatrics with congenital heart diseases due to lower tolerability and reserve capacity and some of them may already have a degree of heart failure. Fluid overload increases the incidence of morbidity and mortality in such patients.

The aim of our study is to observe the amount of fluids needed for flushing during pediatric cardiac catheterization (in ml/kg) and asses its effect on total lung water and PaO2/FiO2, aiming to develop a useful protocol for the amount of fluids used.

DETAILED DESCRIPTION:
.Objectives: The objective of this study is to assess lung water by comparing the calculated values of lung score by ultrasound, PaO2/FiO2 ratio and PaCO2 obtained from arterial blood gases' samples before and after the procedures.

. Study Design:

* A prospective observational study. Study Method
* Population of study & disease condition Children from 1 month to 6 years undergoing cardiac catheterization procedures..
* Study setting:

This study will be conducted at Abo El Reesh Paediatric Hospital, Faculty of Medicine, Cairo University.

- Methodology in details: General anesthesia After interviewing and taking proper history from the parents, examining the patients, checking all routine investigations, informed consent will be taken after discussion with them.

Standard monitoris will be applied to all patients (electrocardiography, pulse oximetry, end-tidal Carbon dioxide CO2, non-invasive arterial blood pressure). All patients will be induced with inhalational induction using 4% sevoflurane in 100% oxygen followed by placement of a peripheral intravenous cannula. Oral endotracheal intubation will be facilitated by IV administration of fentanyl (1-2mic/kg) and atracurium (0.5mg/kg).

Mechanical ventilation will be maintained with an inspired oxygen fraction (FiO2) of 50%, a positive end expiratory pressure (PEEP) of 5 cmH2O, I:E ratio of 1:2 and a peak inspiratory pressure (PIP) will be set to deliver a tidal volume of 5-8 ml/kg and respiratory rate from 15 to 35 cycle per minute according to the end tidal carbon dioxide CO2.

After maintenance of anesthesia and before the procedure lung ultrasound examination will be performed using curved transducer with low frequency (2-5MHz) and will be assessed for the presence of B lines. Arterial blood gases will be aspirated. After the end of the procedure and before awakening the patient both arterial blood gases and lung ultrasound examination will be repeated provided that no complications occurred such as spell or hypertensive crisis.

Maintenance requirements of intravenous fluids will be given by crystalloid solution (lactated ringer) calculated by the "4:2:1 rule": 4 ml/kg/h for the first 10 kg of weight, 2 ml/kg/h for the second 10 kg, and 1 ml/kg/h for each remaining kilograms, in addition preoperative fluid deficits will be replaced calculated by multiplying maintenance requirement per hour by number of hours infant has not received oral or intravenous fluids prior to surgery in aliquots of 50% in the first hour and 25% in second and third hours.

The operators will insert intra-vascular sheathes and catheters that will frequently need to be flushed with heparinized solutions to keep them patent. The amount of the infused solutions will be calculated. This amount will be correlated to the lung ultrasound score.

Lung ultrasound The lung ultrasound score (LUS) is obtained by scanning 12-rib interspaces where each hemithorax divided into 6 areas. Each scanning site yields a score denoting the extent of interstitial pulmonary oedema.

Zero is defined as a complete absence of B-lines in the investigated area. When B-lines are few in the scanning site, they can be easily counted. When they are more numerous, they tend to be confluent and it is less easy to clearly enumerate them. To obtain a semi quantification of the sign, we consider the percentage of scanning site obtained by B-lines (i.e, the percentage of the white screen compared to the black screen below the pleural line) and then divided by 10 (i.e, 30% corresponds to about 3 B-lines, 70% corresponds to about 7 B-lines , and so on). This yields lung score in each site.

Scoring system of lung ultrasound:

Four ultrasound aeration patterns were defined as:

Normal aeration (N): Line sliding sign associated with respiratory movement. Moderate loss of lung aeration (B1 lines) : A clear number of multiple visible B-lines with horizontal spacing between adjacent B lines ≤ 7 mm.

Severe loss of lung aeration (B2 lines): Multiple B lines fused together that were difficult to count with horizontal spacing between adjacent B lines ≤ 3 mm.

White lung,pulmonary consolidation (C): Hyperechoic lung tissue, accompanied by dynamic air bronchogram.

LUS will be determined based on four lung ultrasonographs: N = 0, B1 = 1, B2 = 2 , and C = 3. All patients will undergo a lung ultrasound, and each of the 12 lung areas will be examined. The final LUS of the patient will be the sum of each regional ultrasound score (ranging from 0 to 36).

* Intervention:

Diagnostic intervention: After maintenance of anesthesia and before the procedure lung ultrasound examination will be performed and will be assessed for the presence of B lines. Arterial blood gases will be aspirated. After the end of the procedure and before awakening the patient both arterial blood gases and lung ultrasound examination will be repeated provided that no complications occurred such as spell or hypertensive crisis.

- Potential risks: No additional risks to the study and any risk is related to the surgical procedure itself.

Statistical analysis The Statistical Package of Social Science software program (SPSS), version 21 (Chicago, USA) will be used for all statistical comparisons. Continuous quantitative normally distributed data will be expressed as means and standard deviations (SD), while non-normally distributed data will be expressed as median and range. Qualitative nominal data will be expressed by percentage.

After testing for normality, continuous variables will be compared using t-test or Mann-Whitney U test as appropriate. Categorical variables will be compared using Chi- squared test or Fisher's exact test as appropriate. Changes over time will be compared using ANOVA for repeated measures with Bonferroni correction. Correlation between amount of fluids and lung score will be conducted by pearson's or spearman's methods according to the normality of data. A p-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients undergoing diagnostic cardiac catheterization procedures.

Exclusion Criteria:

* Age <1 month and >6 years.
* Preoperative mechanical ventilation.
* Heart failure
* Patients with oligemic lung diseases.

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children from 1 month to 6 years undergoing cardiac catheterization procedures..
  This study will be conducted at Abo El Reesh Paediatric Hospital, Faculty of Medicine
Sampling Method: Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-10-15 (Estimated); Study Completion 2021-03-15 (Estimated)

PRIMARY OUTCOMES:
Change between lung ultrasound score before and after fluids flushed | at the start of the procedure of cardiac catherization and immediately after the end of the procedure
  heparinized fluids are flushed throughout catheterization through venous and arterial sheathes , ultrasound score will be measured before and after the flushing

SECONDARY OUTCOMES:
. Change between PaO2/FiO2 ratio | immediately before and immediately after the procedure.
  change in ratio between arterial Oxygen tension and Fraction of inspired Oxygen
Correlation between lung score and PaO2/FiO2 ratio | immediately before and immediately after the procedure.
  statistically measuring if there is a relation between lung ultrasound score and PaO2/FiO2 ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Pediatric Hospitals, Giza, الجيزة, Egypt

IPD SHARING:
Plan to Share IPD: Undecided